CLINICAL TRIAL: NCT05153798
Title: Evaluation of PerioMonitor for Detection of Oral Inflammatory Load (OIL) in Human Subjects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oral Science International Inc. (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00055087
Record Dates: First submitted 2021-12-08; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Periodontal Diseases
Keywords: Periodontal; Inflammation; Gingivits; PerioMonitor; Bleeding on Probing; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Inflammation; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PerioMonitor Testing: 117 Subject to be tested for Oral Inflammatory Load (OIL) with PerioMonitor. Same subjects to be tested for Oral Inflammation with the BOP method.

SUMMARY:
The purpose of this multicenter, prospective, single arm Study is to evaluate the efficacy and safety of PerioMonitor as an aid to the presumptive detection of oral inflammation associated with periodontal diseases.

PerioMonitor is an IVD device for the rapid, semi-quantitative detection of PMN in oral samples. This test is intended for prescription use at Point-of-Care ("POC") settings by health care professionals.

DETAILED DESCRIPTION:
PerioMonitor is an IVD device for the rapid, semi-quantitative detection of PMN in oral samples. This test is intended for prescription use at POC settings by health care professionals. This type of In vitro diagnostic device (IVDD) is also sometimes defined as a "Near-Patient Testing" IVDD.

Conducting investigational testing is a pre-requisite to obtain a Class III medical device licence in respect to in vitro diagnostic devices intended for use in POC settings (e.g., home use or outpatient dental clinic) from Health Canada. Such studies are mandatory to establish the safety and effectiveness of the device should be presented to support the performance for each claimed indication for use. They must be conducted on the device using human subjects representative of the intended users and under conditions similar to the conditions of use, to provide reasonable assurance of safety and effectiveness for the intended use. This notably includes:

1. studies to evaluate the sensitivity and the specificity of the device to provide clinically meaningful results in the target population; and
2. consumer fields evaluations, i.e., studies evaluating the performance of the device when used by the intended users without assistance, following instructions provided in the labelling.

The same is also applicable in the United States of America. More specifically with respect to consumer field evaluations, FDA requires clinical data to determine whether particular tests are "simple" and have "an insignificant risk of an erroneous result" to be approved for waiver under the CLIA criteria and cleared for use in POC settings.

This document is a clinical investigational plan specifically designed for the conduct of a blinded, multicenter and prospective, single arm human Study to evaluate the safety and the efficacy of PerioMonitor as an aid to the presumptive detection of oral inflammation associated with periodontal diseases.

This single-arm Study is designed to be representative of the intended use of PerioMonitor as well as the intended users, intended patient population and intended environment of use. To this end, the Study will include a minimum of 117 subjects, tested by HCPs working in three different dental clinics (i.e., with the background, education, and training of those who will perform the test in its intended environment) that are not qualified laboratory technicians, with PerioMonitor.

ELIGIBILITY:
Inclusion Criteria:

* subject > 18 years old;
* subject fluent in English; and
* subject has signed an ICF.

Exclusion Criteria:

* Subject with altered mental status/inability to provide informed consent or follow the procedure of the Study; and
* Previous enrolment into the current Study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected amongst patients visiting the Sites for their scheduled regular exams, which are all outpatient dental clinics
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2021-11-29 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of PerioMonitor | 6 months
  The primary objective of this blinded, multicenter and prospective Study is to evaluate the sensitivity and the specificity of PerioMonitor for semi-quantitative detection of PMN in human oral specimens, which may improve the detection of oral inflammation associated with periodontal diseases. Based on our preliminary results, a sensitivity of 90% (95CI 80.0-100%) and a specificity of 75% (65.1-100%) are expected when testing a cohort of 117 subjects.

SECONDARY OUTCOMES:
Usability of PerioMonitor in Point-of-Care (POC) settings | 6 months
  The secondary objective is to validate the claim that PerioMonitor can be used in POC settings (i.e., representative of the intended users and under conditions similar to the conditions of use), at the time of the consultation, with instant availability of results, by HCPs working in a dental clinic (i.e. with the background, education, and training of those who will perform the test in its intended environment) that are not qualified laboratory technicians, to make immediate and informed decisions about patient care, with a negligible likelihood of erroneous results.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Fort Lee Dental Office, Fort Lee, New Jersey
  - Robert A. Lowe Dental Office, Charlotte, North Carolina
- OMG Perio, Hamilton, Ontario, Canada